CLINICAL TRIAL: NCT06861582
Title: Effect of Point-of-care Analysis of Ultrasensitive Troponin I on Length of Hospital Stay in Patients With Cardiac Chest Pain: a Randomized Study (POC Troponina)
Brief Title: Effect of Point-of-care Analysis of Ultrasensitive Troponin I on Length of Hospital Stay in Patients With Cardiac Chest Pain (POC Troponina)
Acronym: POC Troponina
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ludhmila Abrahão Hajjar MD, PhD, Full Professor of Emergency Medicine, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 83553824.1.0000.0068
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Acute Coronary Syndromes (ACS); Troponin I; Point-of-Care Testing
Keywords: Acute Coronary Syndrome; Non-ST Elevation Myocardial Infarction; Troponin I; Point-of-Care Testing; Biomarkers; Emergency Service, Hospital; Myocardial Ischemia; Cardiovascular Diseases; Hospital Length of Stay
MeSH Terms: conditions — Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction; Emergencies; Myocardial Ischemia; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POC Group (Experimental): For patients randomized to the POC group, the Siemens Atellica VTLi kit will be used. This hs-cTnI test employs a two-site sandwich immunoassay, where anti-cTnI antibodies conjugated to paramagnetic particles bind to cTnI. The particles are manipulated by magnetic fields, allowing optical detection. The biomarker concentration is calculated using a calibration curve.
  The primary sample is whole capillary blood, collected by fingertip puncture. Additionally, patients will have venous ultrasensitive troponin collected using the local laboratory.
  Reference values (99th percentile, pg/mL): Women: 18.5 - Men: 27.1.
  The cTnI values between 0 and LoD are reported as <LoD; values above 1250 pg/mL as >1250 pg/mL. Samples will be taken at times 0 and 1 hour. Analysis will follow the manufacturer's guidelines.
  Interventions: Diagnostic Test: Point-of-care ultrasensitive troponin testing
- Control Group (Placebo Comparator): For patients randomized to the ultrasensitive troponin dosing arm using the local laboratory, the ABBOTT Alinity i kit will be used. Samples will be taken at 0 and 1 hour after admission. The sample for this analysis will be collected by venipuncture and should be drawn into serum tubes with a separator (5 mL capacity).
  The Alinity i STAT High Sensitive Troponin-I assay is a chemiluminescence microparticle immunoassay (CMIA) for the quantitative determination of cardiac troponin I (cTnI) in serum and plasma using the Alinity i analyzer. The analysis will be conducted following the manufacturer's instructions. The measurement range of the assay is 10 to 50,000 pg/mL.
  Population reference values (99th percentile, pg/mL):
  Women (21-75 years): 15.6 Men (21-73 years): 34.2
  Interventions: Diagnostic Test: Laboratory-based ultrasensitive troponin testing

INTERVENTIONS:
Diagnostic Test: Point-of-care ultrasensitive troponin testing — For patients randomized to the ultrasensitive troponin dosing arm using point-of-care (POC) technology, the Atellica® VTLi Patient-side Immunoassay Analyzer (Siemens Healthineers) will be used. This high-sensitivity troponin I (hs-cTnI) test utilizes Magnotech® Technology with paramagnetic particles and external magnetic fields, providing rapid results (~8 minutes) using whole capillary blood collected via fingertip puncture, and/or with direct withdrawal from the test tube. Additionally, venous blood samples will be collected for laboratory comparison. The assay measures hs-cTnI within a range of 0-1250 pg/mL, with values <LoD and >1250 pg/mL recorded accordingly. Samples will be collected at 0 and 1 hour. Reference values (99th percentile, pg/mL): Women: 18.5, Men: 27.1. This intervention enables bedside testing, reducing turnaround time compared to standard laboratory assays, facilitating early myocardial infarction diagnosis.
  Other Names: Atellica® VTLi Patient-side Immunoassay Analyzer
  Arms: POC Group
Diagnostic Test: Laboratory-based ultrasensitive troponin testing — For patients randomized to the ultrasensitive troponin dosing arm using the local laboratory, the Alinity™ i STAT High Sensitive Troponin-I assay (Abbott) will be used. Samples will be taken at 0 and 1 hour after admission by venipuncture and collected in 5 mL serum tubes with a separator. This chemiluminescence microparticle immunoassay (CMIA) quantifies cardiac troponin I (cTnI) in serum and plasma using the Alinity™ i analyzer, with a measurement range of 10-50,000 pg/mL. Analysis will follow the manufacturer's instructions. Reference values (99th percentile, pg/mL): Women (21-75 years): 15.6, Men (21-73 years): 34.2.
  Other Names: Alinity™ i STAT High Sensitive Troponin-I assay
  Arms: Control Group

SUMMARY:
This clinical study aims to compare two different methods for measuring high-sensitivity troponin I, a key biomarker used to diagnose heart attacks.

The primary research question is: Does the use of the Atellica VTLi kit from Siemens for high-sensitivity troponin I (hs-cTnI) testing at the point of care (POC) significantly reduce the average time from admission to hospital discharge compared to the conventional laboratory methodology using the Alinity i kit from ABBOTT?

Participant will:

* Patients aged ≥ 18 years.
* Patients arriving in the emergency room with symptoms suggestive of ACS, with onset of pain between 3 and 12 hours after arrival, in whom serial troponin dosing is planned for investigation.
* Signature of the Informed Consent Form (ICF).

Researchers will analyze whether the point-of-care testing method helps speed up the hospital discharge process compared to the standard laboratory approach. They will also compare the accuracy of the test results, the time taken for clinical decisions, and the overall cost-effectiveness of the two methods.

DETAILED DESCRIPTION:
Objective: evaluation of the length of hospital stays for patients with chest pain in the Emergency Unit of the Heart Institute-HCFMUSP, comparing two methods of ultrasensitive troponin I dosage: the Atellica VTLi kit from Siemens, used in the point of care methodology, and the Alinity i kit from ABBOTT, used in the local laboratory. The aim is to compare the time elapsed between admission and discharge in the two groups, seeking to identify possible differences in the efficiency and speed of care provided by each method.

Background: cardiovascular diseases (CVD) continue to be the main cause of mortality and morbidity in patients admitted to the emergency room with chest pain. Among CVDs, ischemic heart disease is the most lethal, accounting for 38% of all CVD deaths in women and 44% in men. Diagnosis in these cases must be rapid and efficient, since the prognosis improves significantly when treatment is started early in patients with ACS.

Study design: randomized, open, comparative and parallel study at a single center.

Sample size: 200 patients

Intervention: eligible patients will be randomized 1:1 into two groups: the POC dosage group and the control group. In both groups, samples will be taken at time zero and after 1 hour.

Primary outcome: Time between admission of a patient with chest pain symptoms to the emergency department of the Heart Institute-HCFMUSP and discharge after diagnosis of Non-ST Elevation Acute Coronary Syndrome (NSTE-ACS)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years.
* Patients arriving in the emergency room with symptoms suggestive of ACS, with onset of pain between 3 and 12 hours after arrival, in whom serial troponin dosing is planned for investigation.
* Signature of the Informed Consent Form (ICF).

Exclusion Criteria:

* Patients presenting with ACS with ST-segment elevation on the 12-lead ECG on arrival at hospital.
* Patients with conditions that interfere with the interpretation of troponin dosage (chronic renal failure, cancer, chronic lung diseases).
* Pregnant or breastfeeding patients.
* Patients already included in other clinical research protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Time between admission of a patient with chest pain symptoms to the emergency department of the Heart Institute-HCFMUSP and discharge after diagnosis of ACS-NSTE. | 30 days
  From emergency department admission to hospital discharge, assessed up to 30 days, depending on clinical evolution and treatment approach.

SECONDARY OUTCOMES:
Differences in ultrasensitive troponin values obtained by the two methods | At the time of randomization (0-hour) and at 1 hour
  The primary assessment of ultrasensitive troponin values will occur from the first blood sample collection (0-hour) to the second collection (1-hour). Additional blood samples may be collected if clinically indicated, but only within the hospitalization period.
Differences between time from admission to diagnosis of NSTE ACS | 30 days
  From emergency department admission to hospital discharge, assessed up to 30 days, depending on clinical evolution and treatment approach.
Compare the time between blood collection and the result for both groups | 4 hours
  The times at which results become available after each blood sample collection will be assessed, up to 4 hours post-collection.
Determine the time to hospital discharge for patients where ACS has been ruled out (normal hs troponin values) | 24 hours
  From emergency department admission to hospital discharge for patients with normal high-sensitivity troponin (hs-cTn) values, assessed up to 24 hours.
Comparing major adverse cardiovascular events (MACE) | 30 days
  From emergency department admission to the occurrence of major adverse cardiovascular events (MACE) during hospitalization, assessed up to 30 days
Comparison of the cost-effectiveness of the two diagnostic methods for ultrasensitive troponin measurement | 30 days
  The cost-effectiveness of the two diagnostic methods will be assessed in US dollars using the Brazilian Public Health database. This database includes standardized costs for procedures, medications, and hospital stays, allowing for a comparative economic evaluation between point-of-care and laboratory-based ultrasensitive troponin testing.

CONTACTS AND LOCATIONS:
Overall Officials: Ludhmila A Hajjar, Professor, Principal Investigator — University of Sao Paulo
Locations (1):
- Instituto do Coração HCFMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leonel T, Ferreira C, Braz R, Paladino F, Silva H, Gomes S, et al. Clinical and Laboratory Validation of the Atellica vTLi Analyzer for Diagnosis of Myocardial Infarction through High Sensitivity Cardiac Troponin I (hs-cTnI) Measurement. In 2024.
- [Background] Leonel T, Mix A, Vivanco P. Comparison of Performance of High Sensitive Troponin I (cTNIH) by Point-of-care (POC) and Automated cTNIH Immunoassays in Patients at Low Risk of Heart Attack in a Chilean Emergency Unit; Impact on Emergency Department Efficiency. In 2024
- [Background] Gunsolus IL, Schulz K, Sandoval Y, Smith SW, Lindgren B, Okeson B, Apple FS. Diagnostic performance of a rapid, novel, whole blood, point of care high-sensitivity cardiac troponin I assay for myocardial infarction. Clin Biochem. 2022 Jul-Aug;105-106:70-74. doi: 10.1016/j.clinbiochem.2022.04.008. Epub 2022 Apr 18. PMID 35447148
- [Background] Morrow DA, Cannon CP, Jesse RL, Newby LK, Ravkilde J, Storrow AB, Wu AH, Christenson RH; National Academy of Clinical Biochemistry. National Academy of Clinical Biochemistry Laboratory Medicine Practice Guidelines: Clinical characteristics and utilization of biochemical markers in acute coronary syndromes. Circulation. 2007 Apr 3;115(13):e356-75. doi: 10.1161/CIRCULATIONAHA.107.182882. Epub 2007 Mar 23. No abstract available. PMID 17384331
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25. No abstract available. PMID 30153967
- [Background] DeVon HA, Hogan N, Ochs AL, Shapiro M. Time to treatment for acute coronary syndromes: the cost of indecision. J Cardiovasc Nurs. 2010 Mar-Apr;25(2):106-14. doi: 10.1097/JCN.0b013e3181bb14a0. PMID 20142752
- [Background] Than M, Cullen L, Reid CM, Lim SH, Aldous S, Ardagh MW, Peacock WF, Parsonage WA, Ho HF, Ko HF, Kasliwal RR, Bansal M, Soerianata S, Hu D, Ding R, Hua Q, Seok-Min K, Sritara P, Sae-Lee R, Chiu TF, Tsai KC, Chu FY, Chen WK, Chang WH, Flaws DF, George PM, Richards AM. A 2-h diagnostic protocol to assess patients with chest pain symptoms in the Asia-Pacific region (ASPECT): a prospective observational validation study. Lancet. 2011 Mar 26;377(9771):1077-84. doi: 10.1016/S0140-6736(11)60310-3. PMID 21435709
- [Background] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J. 2023 Oct 12;44(38):3720-3826. doi: 10.1093/eurheartj/ehad191. No abstract available. PMID 37622654
- [Background] Writing Committee; Kontos MC, de Lemos JA, Deitelzweig SB, Diercks DB, Gore MO, Hess EP, McCarthy CP, McCord JK, Musey PI Jr, Villines TC, Wright LJ. 2022 ACC Expert Consensus Decision Pathway on the Evaluation and Disposition of Acute Chest Pain in the Emergency Department: A Report of the American College of Cardiology Solution Set Oversight Committee. J Am Coll Cardiol. 2022 Nov 15;80(20):1925-1960. doi: 10.1016/j.jacc.2022.08.750. Epub 2022 Oct 11. No abstract available. PMID 36241466
- [Background] Hsia RY, Hale Z, Tabas JA. A National Study of the Prevalence of Life-Threatening Diagnoses in Patients With Chest Pain. JAMA Intern Med. 2016 Jul 1;176(7):1029-32. doi: 10.1001/jamainternmed.2016.2498. No abstract available. PMID 27295579
- [Background] Mueller C, Giannitsis E, Christ M, Ordonez-Llanos J, deFilippi C, McCord J, Body R, Panteghini M, Jernberg T, Plebani M, Verschuren F, French J, Christenson R, Weiser S, Bendig G, Dilba P, Lindahl B; TRAPID-AMI Investigators. Multicenter Evaluation of a 0-Hour/1-Hour Algorithm in the Diagnosis of Myocardial Infarction With High-Sensitivity Cardiac Troponin T. Ann Emerg Med. 2016 Jul;68(1):76-87.e4. doi: 10.1016/j.annemergmed.2015.11.013. Epub 2016 Jan 12. PMID 26794254
- [Background] Sun BC, Hsia RY, Weiss RE, Zingmond D, Liang LJ, Han W, McCreath H, Asch SM. Effect of emergency department crowding on outcomes of admitted patients. Ann Emerg Med. 2013 Jun;61(6):605-611.e6. doi: 10.1016/j.annemergmed.2012.10.026. Epub 2012 Dec 6. PMID 23218508
- [Background] Gulati M, Levy PD, Mukherjee D, Amsterdam E, Bhatt DL, Birtcher KK, Blankstein R, Boyd J, Bullock-Palmer RP, Conejo T, Diercks DB, Gentile F, Greenwood JP, Hess EP, Hollenberg SM, Jaber WA, Jneid H, Joglar JA, Morrow DA, O'Connor RE, Ross MA, Shaw LJ. 2021 AHA/ACC/ASE/CHEST/SAEM/SCCT/SCMR Guideline for the Evaluation and Diagnosis of Chest Pain: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2021 Nov 30;144(22):e368-e454. doi: 10.1161/CIR.0000000000001029. Epub 2021 Oct 28. PMID 34709879
- [Background] Timmis A, Vardas P, Townsend N, Torbica A, Katus H, De Smedt D, Gale CP, Maggioni AP, Petersen SE, Huculeci R, Kazakiewicz D, de Benito Rubio V, Ignatiuk B, Raisi-Estabragh Z, Pawlak A, Karagiannidis E, Treskes R, Gaita D, Beltrame JF, McConnachie A, Bardinet I, Graham I, Flather M, Elliott P, Mossialos EA, Weidinger F, Achenbach S; Atlas Writing Group, European Society of Cardiology. European Society of Cardiology: cardiovascular disease statistics 2021. Eur Heart J. 2022 Feb 22;43(8):716-799. doi: 10.1093/eurheartj/ehab892. PMID 35016208